CLINICAL TRIAL: NCT04251455
Title: Tissue and Clinical Characterisation of Temporomandibular Joint Diseases
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Bergen (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Bodil Lund, Professor, Karolinska Institutet
Other Study IDs: 2014/622-31/1
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Arthritis; Temporomandibular Joint Disc Displacement; Temporomandibular Joint Osteoarthritis
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthroscopy; Diskectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial tissue: biopsies taken from the superior aspect of the posterior band of the TMJ disc attachment.
  Synovial fluid: synovial fluid samples will be taken with the push-and-pull method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMJ disease/disorder characterisation: Patients with the diagnosis disc displacement without reduction (DDwoR), or disc displacement with reduction (DDwR), or osteoarthritis (OA), or chronic inflammatory arthritis (CIA) were designated to TMJ surgery. According to the Swedish national guidelines on TMJ surgery DDwoR, OA, and CIA patients had arthroscopy and DDwR had discectomy.
  Interventions: Procedure: Arthroscopy or discectomy with sampling of synovial fluid and synovial tissue

INTERVENTIONS:
Procedure: Arthroscopy or discectomy with sampling of synovial fluid and synovial tissue — Arthroscopic lysis and lavage: performed under general anaesthesia. Before initiation of arthroscopy synovial fluid was sampled with a push-and-pull method. The TMJ was investigated with an arthroscope during irrigation with sterile saline solution. Adhesions were addressed with a coblator. Synovial tissue biopsies were taken from the posterior attachment of the disc.
  Discectomy without replacement: performed under general anaesthesia. Before initiation of surgery, synovial fluid was sampled as above described. During surgery synovial tissue biopsies were taken as described above.

SUMMARY:
Temporomandibular joint (TMJ) diseases or dysfunctions affects many patients. Surgical treatment is planned when non-invasive interventions have failed. Still, much is not known regarding aetiology of TMJ diseases and how and why the disease develops over time. The study aims to investigate synovial tissue, synovial fluid and clinical characteristics for patients with TMJ diseases or dysfunctions designated for surgery. Patient samples and clinical variables will be analysed in relation to TMJ diagnosis and related to surgical outcome. The study is a cohort observational study.

DETAILED DESCRIPTION:
TMJ disc displacement is common, affecting 20-30% of the population. Some of these patients will eventually need health-care attention. Patients with TMJ osteoarthritis (OA) or chronic inflammatory arthritis (CIA) are not that common, prevalence numbers are lacking. These TMJ diseases or dysfunctions can severely affect the patients' well-being because of local pain, chewing problems, psychosocial impact, amongst others. Treatment is primarily non-invasive to its character where orthotic splint, physiotherapy, medication, or other treatments can be evaluated. Patients who do not respond to these efforts might have surgery. Arthroscopy is a minimal invasive intervention with a described success rate from 50-90%. From the patients', the society and the surgeons' point of view, better individual pre-operative prognostication is valuable. TMJ disc displacement, OA and CIA is not fully characterised in terms of aetiopathogenesis. There are studies investigating components of extra cellular matrix and cytokines TMJ. The multitude of proteins still not studied may contribute in an unknown fashion to new insights in aetiology and to new treatment opportunities. The aim of the study is to characterise synovial tissue, synovial fluid, and clinical parameters and relate them to the specific TMJ diagnosis but also to each others. A secondary aim is to relate the outcome of surgery to both clinical and tissue variables in order to determine if there are factors that might function as predictors of outcome. A tertiary aim is to investigate if patients who suddenly develops disc displacement without reduction (DDwoR) without any prior signs or symptoms from the TMJ differs in their tissue or clinical characteristics compared to patients who develops DDwoR after having prior signs or symptoms from the TMJ.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* diagnosis DDwoR, DDwR, OA, or CIA
* conservative treatment (i.e. orthotic split, physiotherapy, medication) tried for at least 3-6 months without success

Exclusion Criteria:

* earlier TMJ surgery
* age under 18 years
* patients not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the department of Craniofacial Diseases, Karolinska University Hospital, Stockholm, Sweden, because of disc displacement with reduction (DDwR), disc displacement without reduction (DDwoR), osteoarthritis, and chronic inflammatory arthritis (CIA) were eligible for inclusion. Written informed consent were mandatory. Diagnoses were set according to the Diagnostic Criteria for Temporomandibular Disorders accept CIA, where a rheumatologist had to set the diagnosis. Apart from above mentioned diagnoses criteria for surgery were: visual analogue scale (VAS) value of ≥ 4 for TMJ pain or TMJ disability, and DDwoR patients had to have a maximal interincisal opening (MIO) of ≤ 35 mm.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Characterisation of synovial tissue | 1-5 years after study completion
  Synovial tissue, harvested during surgery, will be assessed through: common histo-pathology analysis, immunohistochemistry, protein analysis in immunoassays, cell characterisation with flow cytometry, and gene expression profiles with PCR.
Characterisation of synovial fluid | 1-5 years after study completion
  Synovial fluid, harvested during surgery, will be assessed through: immunoassays, masspectrometry.

SECONDARY OUTCOMES:
Comparison of protein content | 1-5 years after study completion
  Extracted synovial fluid and synovial tissue will be compared with each other according to protein content.
Outcome of surgery, change in four different variables | Pre-surgery,6 months after surgery
  Outcome of surgery is based on four different variables: objective measurement of MIO (≥35mm), TMJ pain (≤3 on a 0-10 scale), TMJ disability (≤3 on a 0-10 scale), and TMJ psychosocial impact (≤3 on a 0-10 scale). The variables are measured berfore surgery and 6 months after surgery.
Factors predicting surgery | Pre-surgery, during surgery
  Clinical parameters (anamnestic variables,medical variables, TMJ diagnoses and subdiagnoses, objective and subjective measurements) will be related to surgical outcome. Synovial tissue and synovial fluid characteristics (as analysed per above described) related to outcome of surgery.
General joint hypermobility | Pre-surgery.
  Joint mobility measured by the Beighton score, 0-3=normal joint mobility, 4-9 general joint mobility. Joint mobility (general and normal) related to surgical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Lund, Professor, Principal Investigator — Karolinska Institutet, University of Bergen
Locations (1):
- Karolinska Institutet, Department of Dental Medicine, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No